CLINICAL TRIAL: NCT00722969
Title: A Phase II Study of Erlotinib and Sorafenib in Patients With Locally Advanced and/or Metastatic (Stage IIIb or IV) Non Small Cell Lung Cancer Who Have Not Received Prior Chemotherapy
Brief Title: Erlotinib and Sorafenib in Chemonaive Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Free University Medical Center (Other)
Responsible Party: Prof Dr E.F. smit, VU University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07/203; EudraCT: 2007-004625-14
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; erlotinib; sorafenib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: sorafenib + erlotinib

INTERVENTIONS:
Drug: sorafenib + erlotinib — sorafenib 400mg b.i.d oral Erlotinib 150 mg o.i.d oral
  Other Names: nexavar; tarceva

SUMMARY:
Patients with advanced or metastatic (stage IIIB-IV) non small cell lung cancer who have not received prior chemotherapy will be treated with erlotinib 150 mg once a day and sorafenib 400 mg twice a day. The objectives of the study are to assess the efficacy and safety of this combination treatment. Additional exploratory study objectives are correlation of biomarkers and imaging modalities potentially predictive for response and (progression free) survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically advanced NSCLC stage IIIB or IV
2. No prior chemotherapy or therapy with systemic anti-tumor therapy (e.g., monoclonal antibody therapy) or prior exposure to agents directed at the HER axis (e.g. EGFR TK inhibitors, Herceptin). Prior surgery and/or localized irradiation is permitted provided that the irradiated lesion is not the only measurable lesion.
3. Age > 18 years.
4. ECOG Performance Status of 0 or 1
5. Life expectancy of at least 12 weeks.
6. Subjects with at least one uni-dimensional(for RECIST) measurable lesion. Lesions must be measured by CT-scan.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
8. Hemoglobin > 9.0 g/dl
9. Absolute neutrophil count (ANC) >1,500/mm3
10. Platelet count > 100,000/μl
11. Total bilirubin < 1.5 times the upper limit of normal
12. ALT and AST < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
13. Alkaline phosphatase < 4 x ULN
14. PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with low molecular weight heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
15. Serum creatinine < 1.5 x upper limit of normal.
16. Written informed consent.

Exclusion Criteria:

Excluded medical conditions:

1. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy( beta blockers or digoxin are permitted) or uncontrolled hypertension.
2. History of HIV infection or chronic hepatitis B or C.
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 1 months from definitive radiotherapy and off steroids):
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
6. History of organ allograft.
7. Patients with evidence or history of bleeding diathesis
8. Patients undergoing renal dialysis
9. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.

Excluded therapies and medications, previous and concomitant:

1. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
2. Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed). Major surgery within 3 weeks of start of study
3. Autologous bone marrow transplant or stem cell rescue within 4 months of study
4. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
5. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
6. Prior exposure to the study drugs.
7. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
8. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
9. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
10. Patients unable to swallow oral medications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-11 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Rate of non-progression at 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Best overall response rate | end of study
Duration of response | End of study
Survival | End of study
Toxicity | Week 1, week 3, week 6, week 9, week 12 then every 6 weeks
Prediction of early response and effects on tumor vascularisation by PET and perfusion CT scans | Baseline, week 3 and week 6
Biomarkers for response (Proteomics, circulating cells, mutational analysis) | Baseline, week 1, week 3 and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Egbert F Smit, Phd, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (4):
- Netherlands (4):
  - VU university medical center, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
  - University Hospital Maastricht, Maastricht